CLINICAL TRIAL: NCT00792324
Title: A Phase III, Double Blind, Mulit-centre, Randomised Placebo Controlled, Pilot Study to Assess the Feasibility of Switching Individuals Receiving Efavirez With Continuing Central Nervous System (CNS) Toxicity to TMC125.
Brief Title: Pilot Study Switching Individuals Receiving EFV With Continuing Central Nervous System Toxicity to TMC125
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Mark Nelson, St Stephens Aids Trust
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SSAT 029
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: HIV
MeSH Terms: interventions — etravirine; efavirenz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Four 100mg Etravirine tablets plus one Efavirenz (EFV) placebo tablet once daily
  Interventions: Drug: Etravirine
- Group 2 (Active Comparator): One 600mg EFV tablet plus four Etravirine placebo tablet tablets once daily
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Etravirine — Four 100mg tablets daily for 12-24 weeks
  Other Names: TMC125; Brand Name: Intelence
  Arms: Group 1
Drug: Efavirenz — One 600mg tablet daily
  Other Names: TMC125; Brand Name: Intelence
  Arms: Group 2

SUMMARY:
The purpose of the study is to examine the effect of switching from an antiretroviral combination that includes efavirenz (Susitiva®), in individuals experiencing efavirenz-related side effects, and replacing this with an investigational HIV medication called Etravirine (TMC125).

The study will primarily investigate the effect of change in medication on your viral load (the levels of the HIV virus in your blood), on immunological parameters (CD4 count), on other safety parameters (such as cholesterol) your side effects and also on your quality of life.

DETAILED DESCRIPTION:
The majority of individuals who commence treatment for HIV in the UK start with a regimen that includes EFV in combination with other antiretrovirals. These regimens are convenient (once daily dosing) and highly efficacious. However EFV has several potential drawbacks including continued CNS toxicity, the potential for teratogenesis and a low barrier to the development of virological resistance. In the past the only alternative NNRTI available was nevirapine which appears to have a lower rate of virological success and is associated with potentially life threatening toxicities including hepatotoxicity and cutaneous toxicity including the Stevens-Johnson syndrome.

Clinically controlled trials frequently reported undesirable nervous system side effects in patients receiving 600 mg EFV with other antiretroviral agents, including dizziness,insomnia, somnolence, impaired concentration and abnormal dreaming. CNS symptoms of moderate to severe intensity were experienced by 19.4% of patients compared to 9.0% of patients receiving control regimens. These symptoms were severe in 2.0% of patients receiving EFV 600 mg daily and in 1.3% of patients receiving control regimens. In clinical studies 2.1% of patients treated with 600 mg of EFV discontinued therapy because of nervous system symptoms.

Nervous system symptoms usually begin during the first one or two days of therapy and often resolve after the first 2 -4 weeks. However in a significant proportion of individuals it continues with an adverse effect on quality of life. CNS toxicity may also worsen drug compliance. In a study of uninfected volunteers, a representative nervous system symptom had a median time to onset of 1 hour post dose and a median duration of 3 hours.

Nervous system symptoms may occur more frequently when EFV is taken concomitantly with meals possibly due to increased EFV plasma. Dosing at bedtime seems to improve the tolerability of these symptoms and can be recommended during the first weeks of therapy and in patients who continue to experience symptoms although this is not always successful and may be associated with vivid or disturbing dreams. Dose reduction or splitting the daily dose has not been shown to provide benefit.

Other adverse events associated with efavirenz include rash (5-26%, usually minor),increased cholesterol (20-40%) and triglycerides (6-11%), diarrhea (3-14%), nausea and hyperglycemia (2-5%). Serious psychiatric adverse events such as precipitation of psychosis, seizure, suicidal ideation, paranoia, mania and aggression have also been associated with use. These are seen in <1% taking EFV and are thought to be more likely in those with a history of mental illness/drug abuse or predisposition to psychological reactions.

TMC125 is a diarylpyrimidine derivative that has proven efficacy against HIV-1 including activity in viral isolates with existing NNRTI signature mutations. Resistance to TMC125 also appears to develop less readily than to EFV and NVP. This has been attributed to its molecular structure. TMC125 has demonstrated safety and efficacy in short term studies in both treatment-naïve and NNRTI-resistant HIV-1 infected patients.

Recently published results from phase 3 trials give further support to these findings with efficacy in reduction of HIV-1-RNA levels seen in patients with substantial NNRTI and PI resistance when treated with TMC125 plus an optimized background.

TMC-125 is generally well tolerated and in particular has lower reported rates of CNS toxicity than EFV. Animal studies have shown a low risk of teratogenesis. The major toxicity of TMC125 has been skin rash which is usually self-limiting. In the repeated dose trials the adverse events (AEs) reported in more than 10% of all subjects were headache, somnolence, diarrhea, flatulence, nausea and vomiting, fatigue, fever, rash,and pruritus. Overall, AEs were mild to moderate in intensity, with no apparent doseresponse relationship. No consistent or clinically relevant changes in electrocardiogram (ECG) or vital signs were observed with single and repeated TMC125 dosing.

TMC125 is a new NNRTI with proven efficacy against HIV-1 with several potential advantages over EFV including no CNS toxicity and a high barrier to the development of resistance. This study aims to investigate whether substitution of EFV with TMC125 leads to improvement of CNS toxicity with continued virological suppression and immunological reconstitution and whether this is associated with an improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Willing to comply with the protocol requirements
* Has an HIV-plasma viral load at screening <50 HIV-1 RNA copies/mL
* Has a CD4 cell count at screening >50 cells/mm3
* Has been on a stable ART, with at least 3 licensed agents, one of which being EFV, for at least 12 weeks at screening, and is willing to stay on treatment until baseline
* Symptomatic toxicity associated with the EFV after at least 12 weeks of therapy
* If subject is female of childbearing potential, she is using effective birth control methods and is willing to continue practicing these birth control methods during the trial and for at least 30 days after the end of the trial (or after last intake of investigational ARV's)
* If the subject is a heterosexually active male, he is using effective birth control methods and is willing to continue practicing these birth control methods during the trial and until 30 days after the end of the trial (or after the last intake of investigational ARVs)

Exclusion Criteria:

* Subject has a primary HIV-1 infection
* Subject has an HIV-2 infection
* Subject is using any concomitant therapy disallowed by the protocol (as per SPC for EFV and TMC125)
* Subject has any condition (including but not limited to alcohol and drug use) which, in the opinion of the investigator, could compromise the subject's safety or adherence to the protocol
* Subject's life expectancy less than 6 months according to the judgment of the investigator
* subject has a currently active AIDS defining illness (Category C conditions according to the Center for Disease Control [CDC] Classification System for HIV Infection 1993) with the following exceptions, which must be discussed with the sponsor prior to enrollment:
* Stable cutaneous Kaposi's Sarcoma (i.e., no pulmonary or gastrointestinal involvement other than oral lesions) that is unlikely to require any form of systemic therapy during the trial period
* Wasting syndrome due to HIV infection Note: Primary and secondary prophylaxis for an AIDS defining illness is allowed if the medication used is not part of the disallowed medication
* Subject has any active clinically significant disease (e.g., pancreatic, cardiac dysfunction) or findings during Screening of medical history or physical examination that, in the investigator's opinion, would compromise the outcome of the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The rate of neuropsychiatric and central nervous system (CNS) toxicity as measured by the proportion of patients experiencing grade 2-4 neuropsychiatric and CNS toxicity after 12 weeks (as defined by the ACTG adverse event scale). | 12 weeks

SECONDARY OUTCOMES:
The rate of neuropsychiatric and central nervous system (CNS) toxicity after 12 and 24 weeks as measured by the change from baseline by the Hospital Anxiety and Depression Scale (HADS). | 12-24 weeks
Proportion of patients with viral load below 50 copies/mL at weeks 12 and 24 | 12-24 weeks
Proportion of patients with viral load below 400 copies/mL at weeks 12 and 24 | 12 and 24 weeks
Change from baseline in CD4+ count at weeks 12 and 24 | 12 and 24 weeks
Change from baseline in laboratory parameters at weeks 12 and 24 | 12 and 24 weeks
Proportion of patients with non-CNS adverse events at weeks 12 and 24 | 12 and 24 weeks
Change from baseline in adherence at weeks 12 and 24 as measured by the adherence questionnaire: Medication Adherence Self- Report Inventory (M-MASRI) | 12 and 24 weeks
Change from baseline in patient-perceived distress associated with tolerability problems at weeks 12 and 24 as determined by tolerability index questionnaire (HIV patients symptoms profile) | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom